CLINICAL TRIAL: NCT00071097
Title: A Phase II Randomized, Controlled, Partially Blinded Trial to Investigate Dose Response of TMC114/RTV in 3-class-experienced HIV-1 Infected Patients, Followed by an Open-label Period on the Recommended Dose of TMC114/RTV.
Brief Title: TMC114-C202: A Study of Safety, Efficacy, and Tolerability of TMC114 and Low Dose Ritonavir in HIV-1 Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR006778; TMC114-C202; NCT00980928 (obsolete NCT alias)
Record Dates: First submitted 2003-10-10; First posted 2003-10-15 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: HIV Infections
Keywords: HIV; TMC114; Ritonavir; Tolerability; Safety and efficacy; TMC114-C211
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 001 (Experimental): TMC114/rtv 400mg TMC114/100mg rtv once daily
  Interventions: Drug: TMC114/rtv
- 005 (No Intervention): Control Group Control Group, no intervention
- 004 (Experimental): TMC114/rtv 600mg TMC114/100mg rtv twice daily
  Interventions: Drug: TMC114/rtv
- 003 (Experimental): TMC114/rtv 400mg TMC114/100mg rtv both twice daily
  Interventions: Drug: TMC114/rtv
- 002 (Experimental): TMC114/rtv 800mg TMC114/100mg rtv once daily
  Interventions: Drug: TMC114/rtv

INTERVENTIONS:
Drug: TMC114/rtv — 800mg TMC114/100mg rtv once daily
  Arms: 002
Drug: TMC114/rtv — 400mg TMC114/100mg rtv both twice daily
  Arms: 003
Drug: TMC114/rtv — 400mg TMC114/100mg rtv once daily
  Arms: 001
Drug: TMC114/rtv — 600mg TMC114/100mg rtv twice daily
  Arms: 004

SUMMARY:
The purpose of this study is to determine the effectiveness, safety, and tolerability (how well the body stands the drug) of an investigational protease inhibitor (PI) called TMC114 given with low dose ritonavir.

DETAILED DESCRIPTION:
A phase II randomized, controlled, partially blinded, trial to investigate dose response of TMC114/RTV in HIV-1 infected patients who have previously received all three licensed classes of HIV antiviral drugs (known as nucleoside reverse transcriptase inhibitors (NRTI), nonnucleoside reverse transcriptase inhibitors (NNRTI) and protease inhibitors (PI)), and who are on a stable PI-containing regimen not including an NNRTI may be eligible to participate. Four doses of TMC-114/ritonavir will be studied. 300 patients in the United States and Puerto Rico will participate. The duration of the study is 96 weeks. Randomize to one of 4 treatment groups (TMC114/RTV: 400/100 mg qd; 800/100mg qd; 400/100mg bid; 600/100 bid) or control arm for 24 to 48 wks. Optimal dose (TMC114/RTV 600/100mg bid) open label portion of the study. The trial was extended to include 144Wks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older
* Documented HIV-1 infection
* Stable PI regimen for at least 8 weeks prior to screening
* Plasma viral load at screening above 1000 HIV-1 RNA copies/ml
* Prior use of more than 1 NRTI for at least 3 months
* Prior use of one or more NNRTIs as part of a failing regimen
* At least 1 primary PI mutation as defined by the IAS guidelines
* Treatment with at least 1 PI for a total of at least 3 months
* Patient has given informed consent

Exclusion Criteria:

* Presence of any currently active AIDS defining illness except stable cutaneous Kaposi's Sarcoma and Wasting syndrome due to HIV infection
* Current or past history of alcohol and/or drug abuse which, in the investigator's opinion, would compromise the subject's safety or compliance to the study protocol procedures
* NNRTI as part of therapy at screening
* Patients on a treatment interruption at screening
* Patients for whom an investigational antiretroviral therapy is part of the regimen at screening or the use of any non-antiretroviral investigational agents 90 days prior to screening
* Hepatitis A, B, or C.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2003-10; Primary Completion 2005-02 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the dose-response relationship of antiviral activity of the TMC114/RTV dose regimens at 24 Wks in order to determine the optimal dose. | 24 weeks

SECONDARY OUTCOMES:
To evaluate safety and tolerability over 24 to 144Wks; The durability of the antiviral activity; The effect of functional monotherapy with TMC114 over 2 weeks in different doses; and The dose-response by comparing the different TMC114/RTV dosages. | 144 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (39):
- United States (38):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Beverly Hills, California
  - Long Beach, California
  - Los Angeles, California
  - Oakland, California
  - San Diego, California
  - San Francisco, California
  - West Hollywood, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Altamonte Springs, Florida
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Macon, Georgia
  - Chicago, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Camden, New Jersey
  - Albany, New York
  - New York, New York
  - Huntersville, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Dallas, Texas
  - Galveston, Texas
  - Houston, Texas
  - Hampton, Virginia
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Buenos Aires, Argentina

REFERENCES:
- [Result] Clotet B, Bellos N, Molina JM, Cooper D, Goffard JC, Lazzarin A, Wohrmann A, Katlama C, Wilkin T, Haubrich R, Cohen C, Farthing C, Jayaweera D, Markowitz M, Ruane P, Spinosa-Guzman S, Lefebvre E; POWER 1 and 2 study groups. Efficacy and safety of darunavir-ritonavir at week 48 in treatment-experienced patients with HIV-1 infection in POWER 1 and 2: a pooled subgroup analysis of data from two randomised trials. Lancet. 2007 Apr 7;369(9568):1169-78. doi: 10.1016/S0140-6736(07)60497-8. PMID 17416261
- [Derived] De Meyer SM, Spinosa-Guzman S, Vangeneugden TJ, de Bethune MP, Miralles GD. Efficacy of once-daily darunavir/ritonavir 800/100 mg in HIV-infected, treatment-experienced patients with no baseline resistance-associated mutations to darunavir. J Acquir Immune Defic Syndr. 2008 Oct 1;49(2):179-82. doi: 10.1097/QAI.0b013e318183a959. PMID 18769351